CLINICAL TRIAL: NCT02501538
Title: Continuous Diffusion of Oxygen (CDO) Treatment for Healing of Diabetic Foot Ulcers
Acronym: EO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Larry Lavery, Lawrence A Lavery, DPM Study Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 012015-051
Record Dates: First submitted 2015-06-01; First posted 2015-07-17 (Estimated); Results first posted 2020-08-13 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Foot Ulcer, Diabetic
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (1):
- Transcutaneous O2 device (Experimental): Continuous diffusion of oxygen (CDO) (topical oxygen) therapy, which will be administered using a portable device.
  Interventions: Device: Transcutaneous O2 device

INTERVENTIONS:
Device: Transcutaneous O2 device — A portable device that delivers continuous diffusion of oxygen.

SUMMARY:
This is a pilot study. Maximum 30 subjects with a diabetic foot ulcer (DFU) or surgical foot wound will be consented in order to have 20 eligible subjects who will be enrolled and completed the study. Study duration will be three weeks. Patients will be consented and undergo debridement as standard of care at day 0. Ankle-Brachial Index (ABI), Monofilament Sensory Test and Vibration Perception Threshold(VPT) test will be performed only at day 0. Tissue samples will be taken at this visit during standard of care wound debridement and these tissue samples of the wound would normally be removed as part of routine debridement. These tissue samples of the wound will be used for gene expression and bacterial analysis(research). The patient will then receive topical oxygen therapy using the Transcutaneous O2 device (research) with moist wound dressings for 21 days. Moist wound dressings are used as standard of care. Treatment will be initiated during Screening/Baseline visit(day 0) after routine wound debridement, and patient will receive instructions for home use of the device. The patient will be seen for routine wound debridement at days 7, 14, and 21 with a study window of 5 days., Digital photos of the wound, and vascular evaluations (Transcutaneous oxygen measurements and Hyperspectral imaging. will be performed at each study visit(research). Tissue samples will be taken during standard of care wound debridement at every study visit. Results of the data analysis from this project will be used to inform the design of a larger randomized clinical trial.

DETAILED DESCRIPTION:
Patients seen at the University of Texas (UT) Southwestern Wound Clinic with a diabetic foot wound will be identified, consented, and screened for the study. Upon signing consent, patients will be assigned a unique screening number. The screening number given to the first patient will be 01 and increasing sequentially with each subject screened. Screened subjects will be entered onto a screening log. Once a number is assigned it cannot be re-assigned to another subject.

At Day 0, a vascular evaluation including ABI, Sensilase, Transcutaneous oxygen measurements, and hyperspectral imaging will be performed. Monofilament Sensory Test and Vibration Perception Threshold(VPT) test will also be performed at day 0.Patients will undergo standard of care wound debridement. Tissue samples will be taken routinely as standard of care. A wound assessment will be performed, including the debridement as standard of care, wound measurements, and digital photos. Gene expression and bacterial analysis will be performed on tissue samples. After tests are performed, patient will receive topical oxygen therapy using the Transcutaneous O2 device with moist wound dressings. Moist wound dressings are used as standard of care. Patient will receive instructions to continue treatment at home.

Patient will return for an appointment at days 7, 14, and 21, where vascular assessment (Sensilase, Transcutaneous oxygen measurements, Hyperspectral imaging) ,wound assessment (wound measurements, digital photos and acetate tracings) and tissue sampling will be performed following standard of care debridement, Patient will cease topical oxygen treatment at day 21, and study will be concluded.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of all races and ethnicities, age 18-89
* Diagnosis of diabetes mellitus
* Has a diabetic foot ulcer

Exclusion Criteria:

* End-stage renal disease (ESRD)
* Has untreated foot ulcer at time of study
* HIV, hepatitis, autoimmune disease, Systemic lupus erythematous (SLE), Raynaud's disease
* Ankle-Brachial Index (ABI) < 0.4
* Unable or unwilling to provide informed consent

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2020-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A Lavery, DPM, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center at Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transcutaneous O2 Device
Started | 23
Completed | 20
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Transcutaneous O2 Device
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 11
  African American | 5
  Hispanic | 7

OUTCOME MEASURES:

1. Primary Outcome: Tissue Oxygenation as Measured by Hyperspectral Imaging
Description: Hyperspectral (HyperMed, Inc.) images were taken for evaluation of tissue oxygenation following debridement at Visit 1 (day 0), visit 2 (day 7), visit 3 (day 14), visit 4 (day 21). Two images were taken of the study foot - one of the plantar surface and one of the dorsal surface to evaluate the oxygenation of the entire foot. Measurements of oxygenated hemoglobin are generated by the camera for each image. Results are reported in aggregate as mean/standard error for all time points.
Time Frame: 21 days
Population: There was no control arm for this study. For analysis, groups were analyzed as "healer" and "nonhealer." Healers are defined by those patients who achieved a 50% wound area reduction in the study time frame and are likely to heal within 12 weeks. Nonhealers did not reach a 50% wound area reduction in the study time frame.
Measure: Mean (Standard Error); unit: percent concentration of oxyhemoglobin
Arm/Group | Transcutaneous O2 Device
Number analyzed (Participants) | 23
percent concentration of oxyhemoglobin
  Dorsal oxyhemoglobin - healer: number analyzed (Participants) | 12
  Dorsal oxyhemoglobin - healer | 63.58 (11.17)
  Dorsal oxyhemoglobin - nonhealer: number analyzed (Participants) | 11
  Dorsal oxyhemoglobin - nonhealer | 61.91 (9.14)
  Plantar oxyhemoglobin - healer: number analyzed (Participants) | 12
  Plantar oxyhemoglobin - healer | 76.33 (4.86)
  Plantar oxyhemoglobin - nonhealer: number analyzed (Participants) | 11
  Plantar oxyhemoglobin - nonhealer | 77.55 (5.90)

2. Primary Outcome: Tissue Perfusion as Measured by TCPO2
Description: Transcutaneous oxygen pressure (TCPO2) was measured at visit 1 (day 0), visit 2 (day 7), visit 3 (day 14), visit 4 (day 21) to assess perfusion of the tissue. This is measured at the medial and lateral foot to include both major blood vessels to the foot. Reported here as aggregate mean over all time points.
Time Frame: 21 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg
Groups:
- Transcutaneous Oxygen Measurements: Medial and lateral foot measurements
Arm/Group | Transcutaneous Oxygen Measurements
Number analyzed (Participants) | 23
mmHg
  Transcutaneous oxygen - medial foot - healer: number analyzed (Participants) | 12
  Transcutaneous oxygen - medial foot - healer | 53.31 (4.33)
  Transcutaneous oxygen - medial foot - nonhealer: number analyzed (Participants) | 11
  Transcutaneous oxygen - medial foot - nonhealer | 53.64 (3.97)
  Transcutaneous oxygen - lateral foot - healer: number analyzed (Participants) | 12
  Transcutaneous oxygen - lateral foot - healer | 55.21 (3.46)
  Transcutaneous oxygen - lateral foot - nonhealer: number analyzed (Participants) | 11
  Transcutaneous oxygen - lateral foot - nonhealer | 59.31 (4.68)

3. Secondary Outcome: Change in Levels of Growth Factors and Cytokines Involved in Wound Healing
Description: Comparison of measurements inflammatory cytokines: Interleukin 6 (IL-6), Interleukin 8 (IL-8), tumor necrosis factor (TNF)-α and growth factors: vascular endothelial growth factor (VEGF), platelet derived growth factor (PDGF), insulin derived growth factor (IGF), transforming growth factor beta (TGF)-β. These are reported as log fold change by delta delta ct.
  Evaluated from tissue samples obtained at visit 1 (day 0), visit 2 (day 7), visit 3 (day 14), visit 4 (day 21).
Time Frame: 21 days
Measure: Mean (Standard Error); unit: log fold change
Groups:
- Cytokine and Growth Factor Measurement: Measurement of cytokines
Arm/Group | Cytokine and Growth Factor Measurement
Number analyzed (Participants) | 23
log fold change
  IL-6 visit 1 | 2.68 (0.82)
  IL-6 Visit 2 | 11.37 (5.11)
  IL-6 Visit 3 | 18.24 (6.48)
  IL-6 Visit 4 | 9.12 (2.53)
  IL8 visit 1 | 3.97 (1.90)
  IL8 visit 2 | 3.12 (1.31)
  IL8 visit 3 | 7.51 (2.89)
  IL8 visit 4 | 5.22 (2.38)
  TNFa visit 1 | 1.82 (0.41)
  TNFa visit 2 | 8.17 (2.26)
  TNFa visit 3 | 5.03 (1.73)
  TNFa visit 4 | 3.27 (1.19)
  VEGF visit 1 | 1.37 (0.26)
  VEGF visit 2 | 5.85 (1.40)
  VEGF visit 3 | 4.35 (1.42)
  VEGF visit 4 | 3.29 (0.99)
  PDGF visit 1 | 1.40 (0.23)
  PDGF visit 2 | 3.92 (1.31)
  PDGF visit 3 | 1.76 (0.37)
  PDGF visit 4 | 1.81 (0.52)
  IGF1 visit 1 | 3.04 (1.18)
  IGF1 visit 2 | 19.91 (9.10)
  IGF1 visit 3 | 5.47 (2.46)
  IGF1 visit 4 | 5.25 (2.0)
  TGFb visit 1 | 1.27 (0.19)
  TGFb visit 2 | 10.42 (3.05)
  TGFb visit 3 | 4.65 (1.22)
  TGFb visit 4 | 3.96 (1.26)

4. Secondary Outcome: Evaluate Changes in Bacterial Infection
Description: Tissue samples sent for 16s rRNA quantitative culture. Reported in aggregate for each visit that corresponds to Visit 1 (day 0), visit 2 (day 7), visit 3 (day 14), visit 4 (day 21).
Time Frame: 21 days
Measure: Mean (Standard Deviation); unit: CFU/ml
Groups:
- Quantitative Bacterial Cultures: Quantitative bacterial cultures by visit
Arm/Group | Quantitative Bacterial Cultures
Number analyzed (Participants) | 23
CFU/ml
  Visit 1 | 137071.35 (204854.93)
  Visit 2 | 433719.88 (1009663.23)
  Visit 3 | 276842.20 (603627.08)
  Visit 4 | 598557.90 (2303848.45)

5. Secondary Outcome: Percent Wound Area Reduction
Description: Percent change of the wound area (measured in cm^2) of visit 2 (day 7), visit 3 (day 14), and visit 4 (day 21) compared to baseline.
  Percent area reduction = initial surface area (length in cm x width in cm) minus current surface area (length in cm x width in cm), divided by initial surface area. multiplied by 100 to get percentage.
Time Frame: 21 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percent change of wound area (cm^2)
Arm/Group | Transcutaneous O2 Device
Number analyzed (Participants) | 23
percent change of wound area (cm^2)
  Wound area reduction - visit 1 - healers: number analyzed (Participants) | 12
  Wound area reduction - visit 1 - healers | 40.75 (8.26)
  Wound area reduction - visit 3 - healers: number analyzed (Participants) | 12
  Wound area reduction - visit 3 - healers | 48.64 (6.82)
  Wound area reduction - visits 4 - healers: number analyzed (Participants) | 12
  Wound area reduction - visits 4 - healers | 59.91 (7.55)
  Wound area reduction - visit 2 - nonhealers: number analyzed (Participants) | 11
  Wound area reduction - visit 2 - nonhealers | 7.59 (6.32)
  Wound area reduction - visit 3 - nonhealers: number analyzed (Participants) | 11
  Wound area reduction - visit 3 - nonhealers | -30.07 (17.25)
  ound area reduction- visit 4 - nonhealers: number analyzed (Participants) | 11
  ound area reduction- visit 4 - nonhealers | -11.21 (14.50)

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | Transcutaneous O2 Device
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 1/23
Other Adverse Events (participants affected / at risk) | 2/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transcutaneous O2 Device (N=23)
Celluliltis (Skin and subcutaneous tissue disorders) | 1 — Unilateral leg cellulitis, nonstudy leg
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Transcutaneous O2 Device (N=23)
Abrasion (Skin and subcutaneous tissue disorders) | 1 — Abrasion from offloading boot
Foot swelling (Skin and subcutaneous tissue disorders) | 1 — Swelling of study foot

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT02501538/Prot_SAP_ICF_000.pdf